CLINICAL TRIAL: NCT04131023
Title: Metabolic Tracking During Pregnancy to Promote Adequate Gestational Weight Gain
Brief Title: Metabolic Tracking and Weight Gain During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Corrie Whisner, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006557
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Gestational Weight Gain
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metabolic Tracking (Experimental): Metabolism (indirect calorimetry) tracking was performed
  Interventions: Behavioral: Breezing Metabolic Rate Tracking
- Standard Care (No Intervention): Metabolic (indirect calorimetry tracking was not performed

INTERVENTIONS:
Behavioral: Breezing Metabolic Rate Tracking — Metabolism (indirect calorimetry) data were collected every two weeks over 13 weeks of gestation across the second trimester (weeks 13-27) and the values obtained were provided to the participant without health education.
  Arms: Metabolic Tracking

SUMMARY:
In this study, the investigators aimed to have pregnant women use a hand-held device to track increases in daily caloric needs during pregnancy. Weight gain was assessed over time with the goal of reducing excessive gestational weight gain relative to a group of pregnant women who received standard prenatal care.

DETAILED DESCRIPTION:
Specific Aims

The investigators pursued the following specific aims:

1. Evaluate the impact of a mobile, real-time metabolism tracking device on gestational weight gain (GWG) (i.e. total weight gain and rate of weight gain) in pregnant women. The investigators postulated that the metabolism tracking (Breezing) group would have a higher proportion of women who gain the appropriate amount of weight per IOM recommendations. Further, the investigators expected the women in the Breezing group to gain a mean weight within +/- 3 lbs of their recommended GWG range per IOM guidelines, compared to standard care-receiving controls.
2. Assess changes in resting energy expenditure during pregnancy in relation to self-reported dietary intake (at baseline, 4 weeks, 8 weeks, and 12 weeks). The investigators hypothesized that energy requirements would change across the second trimester and that self-reported caloric intakes would correlate with resting energy expenditure (REE)-corrected values (from Breezing) for women in the Breezing group.

Exploratory Aims

1. Evaluate the associations among objective and self-reported sleep parameters (actigraphic total sleep time, sleep onset latency, wake after sleep onset, and mid-sleep point; sleep diary total sleep time, sleep onset latency, wake after sleep onset, and mid-sleep point; insomnia symptoms; and sleep disordered breathing risk) and GWG within the Breezing and control groups.

ELIGIBILITY:
Inclusion Criteria:

* All English and Spanish-speaking, pregnant women
* Gestational age < 17 weeks at time of recruitment
* Aged 18 years or older

Exclusion Criteria:

* High-risk pregnancies that include the following diseases or conditions: fetal growth problems, medical history of hypertension, gastrointestinal disorders, malabsorptive diseases, hyper or hypo-parathyroid conditions, HIV, diabetes (Types 1 and 2 or gestational diabetes), asthma/lung disease, cardiac disease or conditions, current smoker (i.e. women who have smoked 100 cigarettes in their lifetime and now smoke every day or some days) history of eating disorder, or other metabolic conditions known to affect maternal health and fetal development
* Women pregnant with multiple gestations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-17 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Gestational Weight Gain | 0 weeks, 3 weeks, 5 weeks, 7 weeks, 9 weeks, 11 weeks, 13 weeks
  Change in body weight from study baseline to 13 weeks
Change in Resting Energy Expenditure | 0 weeks, 3 weeks, 5 weeks, 7 weeks, 9 weeks, 11 weeks, 13 weeks
  Change in resting energy expenditure, measued by indirect calorimetry, from study baseline to 13 weeks

SECONDARY OUTCOMES:
Change in Total Sleep Time | 0 weeks, 5 weeks, 11 weeks
  Change in total sleep time, measured by wrist-worn actigraphy on the non-dominant arm, from study baseline to 11 weeks
Change in Sleep Onset Latency | 0 weeks, 5 weeks, 11 weeks
  Change in sleep onset latency, measured by wrist-worn actigraphy on the non-dominant arm, from study baseline to 11 weeks
Change in Wake After Sleep Onset | 0 weeks, 5 weeks, 11 weeks
  Change in wake after sleep onset, measured by wrist-worn actigraphy on the non-dominant arm, from study baseline to 11 weeks
Change in Mid-Sleep Point | 0 weeks, 5 weeks, 11 weeks
  Change in mid-sleep point, measured by wrist-worn actigraphy on the non-dominant arm, from study baseline to 11 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No